CLINICAL TRIAL: NCT05759026
Title: The Management of Pain and Anxiety, Using Virtual Reality, During the Care of Elderly Hospitalized Patients
Brief Title: Comparison of the Benefits of a Personalized Intervention (Virtual Environment and Device) Compared to Usual Care
Acronym: ADA-VRSPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-PP-23
Record Dates: First submitted 2023-02-14; First posted 2023-03-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Elderly

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control condition (Experimental): The patient will be randomized so that the kind of intervention will be determined in a random way.
  Interventions: Other: Accompaing cares
- with VR (Experimental): The patient will be randomized so that the kind of intervention will be determined in a random way.
  Interventions: Other: Accompaing cares
- with VR personalised (Experimental): The patient will be randomized so that the kind of intervention will be determined in a random way.
  Interventions: Other: Accompaing cares

INTERVENTIONS:
Other: Accompaing cares — After signing the consent form, the patient will be randomised. The ones randomised in VR groups will choose their preferred environment (e.g. landscapes, animals...).
  The participant will be managed during 1 care (one care in control condition (no material used), care with the VR headset, one care with the VR set and the prefered environnent of the patient) for an average of 30 minutes (including the completion of the scales and questionnaires).

SUMMARY:
The medical environment can create stressful and anxiety-provoking situations for patients, especially during painful procedures, particularly in older adults. These stressful environments have a deleterious effect on the quality of care, even putting the patient at risk and the health care team at risk. The search for a solution is therefore imperative. The evolution of new technologies, such as virtual reality (VR), seems to be an answer to this challenge. Through a multidisciplinary research (psychology and medicine), this project proposes to study the factors allowing to improve the management of older adults during their care using VR. More precisely, different individual factors (age, cognitive level, individual preferences...) and different virtual reality universes (relaxation, landscapes...) on different supports (headsets and touch tablet) will be studied in order to understand the roles of these factors on pain and anxiety management during care procedures. This trial is an interventional, randomized, open-label, single-center study of 100 people over 60 years old. The aim of this project is to improve the quality of life of hospitalized patients but also of caregivers in their work environment. It is expected a significant reduction of pain and anxiety during the intervention with a personalized equipment and environment, compared to usual care conditions. The hypotheisis is also that these interventions, aimed at reducing pain and anxiety in patients, will have beneficial effects on the quality of work life of the caregivers performing the care.

DETAILED DESCRIPTION:
The management of pain and anxiety, during care, will be proposed to patients hospitalized in the geriatric department of the Cimiez Hospital in Nice. After signing the consent form, the equipment and the different virtual environments will be presented to the patient and he will choose his preferred environment.Each patient will be accompanied during a treatment (either in control condition, or in VR condition with a VR condition with a personalised environment (VREP), or in VR condition with a environment (VRNP) for an average of 15 minutes (including the completion of the (including the completion of scales and questionnaires). Assessments will be carried out just before the treatment and just after the treatment.

After the treatment, the caregiver will also be asked to complete a scale assessing After the treatment, the carer will also be asked to complete a scale assessing the treatment (2 minutes on average to complete this scale).

And at the end of the study, the caregivers who participated in the study will be asked to rate their acceptability of VR using the User Experience Survey.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Over 60 years old
* Subject affiliated to the Social Security
* Patient receiving 4 identical cares as part of routine care

Exclusion Criteria:

* Presence of visual and auditory disorders contraindicating the use of a VR headset;
* Unstabilized epilepsy;
* Acute psychiatric disorders
* Vulnerable population

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) - Pain and Anxiety | immediatly before care
  The Visual Analog Scale (VAS) is a self-report scale that allows the patient to evaluate their feelings using a slider that goes from 0 to 10 points (worse score is 10)
Visual Analog Scale (VAS) - Pain and Anxiety | immediatly after care
  The Visual Analog Scale (VAS) is a self-report scale that allows the patient to evaluate their feelings using a slider that goes from 0 to 10 points (worse score is 10)

SECONDARY OUTCOMES:
HAD scale (Hospital Anxiety Depression scale) | immediately beafore care
  This scale evaluates the anxiety that a subject presents, only in a given situation. This tool proposes statements to patients who must then indicate whether their current state corresponds to this statement. The patients can answer from 0 to 3 according to their current feeling. This questionnaire includes 7 items allowing to evaluate the anxiety of the patient. Higher score and worse score: 21
HAD scale (Hospital Anxiety Depression scale) | immediately after care
  This scale evaluates the anxiety that a subject presents, only in a given situation. This tool proposes statements to patients who must then indicate whether their current state corresponds to this statement. The patients can answer from 0 to 3 according to their current feeling. This questionnaire includes 7 items allowing to evaluate the anxiety of the patient. Higher score and worse score : 21
Algo Plus Scale | during care
  The algoplus scale is a scale assessing pain in five categories of behaviors to be observed: face, gaze, complaints, body and general behavior. Only one behavior in a category needs to be observed to be considered active. Each active category, regardless of the number of behaviors observed, counts as one point. This scale evaluates from 0 (minimum score) to 5 (maximum score). The presence of pain is diagnosed if the total score is greater than or equal to 2
Heart rate measurment with Oximeter | 2 minutes before the medicale procedure
  The heart rate is measured with the number of pulses per minute. This measurement aims to evaluate the changes in the heart rate that may be related to an emotional response (positive or negative) related to the care and / or the intervention implemented (VR and / or tablet).
Heart rate measurment with Oximeter | 2 minutes after the medicale procedure
  The heart rate is measured with the number of pulses per minute. This measurement aims to evaluate the changes in the heart rate that may be related to an emotional response (positive or negative) related to the care and / or the intervention implemented (VR and / or tablet).
Respiratory rate with Oximeter | 2 minutes before the medicale procedure
  The respiratory rate is the number of respiratory cycles (inhalation and exhalation) per unit of time, of each individual. This measurement aims to observe changes in the breathing rhythm related to a strong emotion (positive or negative) that could be related to the care and/or the intervention implemented.
Respiratory rate with Oximeter | 2 minutes after the medicale procedure
  The respiratory rate is the number of respiratory cycles (inhalation and exhalation) per unit of time, of each individual. This measurement aims to observe changes in the breathing rhythm related to a strong emotion (positive or negative) that could be related to the care and/or the intervention implemented.
Digital scale of care completion | after each care
  After treatment, a numerical scale will be proposed to the caregiver who performed the treatment, in order to evaluate the performance of the treatment (difficulties, observation of the patient: discomfort/pain, quality of treatment). The associate investigator will then ask the caregiver to rate each item from 0 to 10. Worse outcome : 10
System Usability Scale (SUS) | at the end of the study
  To obtain the SUS score, the contributions to the score of each item must first be added together. The contribution to the score of each item ranges from 1 to 5. For items 1, 3, 5, 7, and 9, the contribution to the score is equal to the position on the scale minus 1. For items 2,4,6,8, and 10, the contribution is 5 minus the position on the scale.Multiply the sum of the scores by 2.5 to get the overall SU value. SUS scores range from 0 to 100. The higher the score, the greater the acceptability and usability

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice - Hopital de Cimiez, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbel C, Le Cerf F, Capriz F, Vaillant-Ciszewicz AJ, Breaud J, Guerin O, Corveleyn X. The management of pain and anxiety using virtual reality during the care of elderly hospitalized patients: Study protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Aug;155:107990. doi: 10.1016/j.cct.2025.107990. Epub 2025 Jun 23. PMID 40562303